CLINICAL TRIAL: NCT05818267
Title: Efficacy and Safety of Regorafenib Maintenance Therapy in Patients With Metastatic Colorectal Cancer (mCRC) Without Imaging Progress Three Months After Second-Line Treatment
Brief Title: Efficacy and Safety of Regorafenib Maintenance Therapy in Patients With Metastatic Colorectal Cancer (mCRC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Zhang (Other)
Responsible Party: Sponsor-Investigator, Wei Zhang, Profrssor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-SUSTAIN
Record Dates: First submitted 2023-02-24; First posted 2023-04-18 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The drug dose that taken by the subject is gradually increased to the maximum dose tolerated by the patient according to individualization. Specifically, the initial dose of 80 mg/day was gradually increased to 120 mg/day (80 mg/day in the first week, 120 mg/day in the second week, and a maximum tolerated dose of 160 mg/day). The maximum tolerated dose is 160 mg/day. The dose is administered once daily in a 4-week cycle (3 weeks of dosing and 1 week of rest) and the maximum dose achieved in the first treatment cycle is maintained.At the discretion of the investigator, regorafenib may be delayed or discontinued. Dose adjustments and interruptions due to toxicity are made according to the recommendations specified in the protocol.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — The drug dose that taken by the subject is gradually increased to the maximum dose tolerated by the patient according to individualization. Specifically, the initial dose of 80 mg/day was gradually increased to 120 mg/day (80 mg/day in the first week, 120 mg/day in the second week, and a maximum tolerated dose of 160 mg/day). The maximum tolerated dose is 160 mg/day. The dose is administered once daily in a 4-week cycle (3 weeks of dosing and 1 week of rest) and the maximum dose achieved in the first treatment cycle is maintained.At the discretion of the investigator, regorafenib may be delayed or discontinued. Dose adjustments and interruptions due to toxicity are made according to the recommendations specified in the protocol.

SUMMARY:
Regorafenib in third-line treatment of metastatic colorectal cancer(mCRC) significantly prolongs the survival of patients, and its advancement has a sensitizing effect on postline chemotherapy and thus improves the prognosis of patients. Therefore, the present study was designed to include patients who achieved stable disease/partial response(SD/PR) after 3 months of second-line therapy and advance regorafenib to investigate the role of advance regorafenib in prolonging progression-free survival, prolonging the efficacy of overall survival, safety, and quality of life in patients with mCRC compared with standard second-line and third-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic colorectal cancer who have measurable metastatic disease according to the Resolute Efficacy Criteria for Solid Tumors (RECIST) version 1.1.
* Received standard second-line therapy, achieved stable disease(SD) and above by recist1.1 tumor assessment and maintained for 3 months.
* Eastern Oncology Collaborative Group(ECOG) physical status of 0 or 1 at trial entry and life expectancy ≥ 3 months.
* No bone marrow suppression and normal heart, lung, liver and kidney function.
* Voluntary participation in research.

Exclusion Criteria:

* Concurrent primary tumors of other types.
* MSI-H/dMMR type mCRC patients.
* Heart, liver, kidney, bone marrow insufficiency or mental abnormalities.
* Intolerant to treatment methods
* Concurrent participants in other clinical trials.
* Pregnant or lactating women.
* Patients deemed unsuitable for study participation by the remaining investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
duration of disease control(DDC) | 6 month
  From second-line treatment initiation to third disease progression

SECONDARY OUTCOMES:
Overall Survival(OS) | 3 years
  Subjects were censored from the time of enrollment to the time of death from any cause, and the date of censoring was the date of the last follow-up visit if the subject's last status was alive.
Quality-of-Life(QoL) | 3 years
  Quality-of-life was evaluated using the Quality-of-Life Questionnaire C30 (EORTC QLQ-C 30) developed by the European organization for research and treatment of cancer (EORTC)
The incidence of adverse events | 3 years
  Adverse Events (AE) will be evaluated and graded according to NCI-CTCAE v5.0. All adverse events will be reported at length.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China